CLINICAL TRIAL: NCT01030133
Title: Effects of TMS and Stimulus Controllability on Pain Perception
Brief Title: Effects of Transcranial Magnetic Stimulation (TMS) and Stimulus Controllability on Pain Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Borckardt_19079
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Chronic Pain
Keywords: Pain
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Real TMS (Active Comparator): Participants in the real Transcranial Magnetic Stimulation (TMS) group will receive real stimulation across all interventions; the operator role Real TMS and receiver role Real TMS. rTMS will be used to stimulate the left prefrontal cortex using two Neuronetics TMS machines with figure-8, iron core coils at 10Hz and at 110% of resting motor threshold [5 second trains following each trial (25 trials per visit)].
  Interventions: Device: Operator Role Real TMS; Device: Receiver Role Real TMS
- Sham TMS (Sham Comparator): Participants in the sham Transcranial Magnetic Stimulation (TMS) group will receive sham stimulation across all interventions; the operator role Sham TMS and receiver role Sham TMS. Sham Stimulation involves 5 second trains of 10Hz rTMS in pairs alternating between real TMS and eSham TMS (randomly ordered). All sham treatment will be delivered with a specially designed, manufacture-provided sham TMS coil that looks and sounds identical to a real TMS coil but no magnetic current is transferred to the participant.
  Interventions: Device: Operator Role Sham TMS; Device: Receiver Role Sham TMS
- All Participants Operator Role (Other): All participants in Operator Role (Receiving real or sham TMS)
  Interventions: Device: Operator Role Real TMS; Device: Operator Role Sham TMS; Device: All Participants Operator Role

INTERVENTIONS:
Device: Operator Role Real TMS — In two of the four visits, the participant will be assigned to the operator condition receiving Real TMS. The participant will be assigned a partner and both participants will participate in a numeric-combination-guessing task. Performance on this task will be directly related to the painfulness of a series of thermal stimuli that participants receive. The "operator's" performance will control the painfulness delivered to both participants. Each participant will play each role twice.
  Arms: All Participants Operator Role; Real TMS
Device: Receiver Role Real TMS — In two of the four visits, the participant will be assigned to the receiver condition receiving Real TMS. The participant will be assigned a partner and both participants will participate in a numeric-combination-guessing task. Performance on this task will be directly related to the painfulness of a series of thermal stimuli that participants receive. The "receiver's" performance on the task will be unrelated to his/her stimulus painfulness. Each participant will play each role twice.
  Arms: Real TMS
Device: Operator Role Sham TMS — In two of the four visits, the participant will be assigned to the operator condition receiving Sham TMS. The participant will be assigned a partner and both participants will participate in a numeric-combination-guessing task. Performance on this task will be directly related to the painfulness of a series of thermal stimuli that participants receive. The "operator's" performance will control the painfulness delivered to both participants. Each participant will play each role twice.
  Arms: All Participants Operator Role; Sham TMS
Device: Receiver Role Sham TMS — In two of the four visits, the participant will be assigned to the receiver condition receiving Sham TMS. The participant will be assigned a partner and both participants will participate in a numeric-combination-guessing task. Performance on this task will be directly related to the painfulness of a series of thermal stimuli that participants receive. The "receiver's" performance on the task will be unrelated to his/her stimulus painfulness. Each participant will play each role twice.
  Arms: Sham TMS
Device: All Participants Operator Role — All participants in Operator Role (Receiving real or sham TMS)
  Arms: All Participants Operator Role

SUMMARY:
Although transcranial magnetic stimulation (TMS) is now considered a minimal risk intervention, is approved for the treatment of depression, and is widely used around the world, little is known about mechanisms of action of prefrontal rTMS for depression or pain. There is some evidence that the prefrontal cortex is involved in perception of control and may moderate the effects of perceived controllability on emotional reactivity to painful stimuli. The present study aims to investigate the effects of prefrontal rTMS and perceived controllability on pain perception in healthy adults.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a minimally invasive brain stimulation technology that can focally stimulate the brain of an awake individual.1,2 A localized pulsed magnetic field transmitted through a figure-8 coil (lasting only microseconds) is able to focally stimulate the cortex by depolarizing superficial neurons3,4 which induces electrical currents in the brain.5 If TMS pulses are delivered repetitively and rhythmically, the process is called repetitive TMS (rTMS).

rTMS over the prefrontal cortex has been shown to produce temporary analgesic effects in healthy adults using laboratory pain methods and in patients with chronic pain of various etiologies. However, little is known about mechanisms of action.

Evidence from functional MRI studies suggests that participants' perceived controllability over pain stimuli is associated with decreased pain experience and decreased activation of cortical and subcortical areas involved with pain perception.6 Perceived controllability may involved prefrontal cortical circuits and may be involved in inhibition of limbic system responses to painful stimuli.

To date, no studies have investigated the interaction between prefrontal TMS and perceived controllability on pain perception in healthy adults. Building on extensive pilot work and experience in the area of laboratory pain assessment and TMS in the Brain Stimulation Laboratory at MUSC, the investigators propose to investigate the effects of perceived controllability and prefrontal TMS on pain perception in healthy adults. This study may help determine whether TMS can be used to stimulate a cortical area thought to be involved in perceived controllability, thus enhancing one's sense of controllability and thereby substantially reduce pain intensity and unpleasantness.

Although transcranial magnetic stimulation (TMS) is now considered a minimal risk intervention, is approved for the treatment of depression, and is widely used around the world, little is known about mechanisms of action of prefrontal rTMS for depression or pain. There is some evidence that the prefrontal cortex is involved in perception of control and may moderate the effects of perceived controllability on emotional reactivity to painful stimuli. The present study aims to investigate the effects of prefrontal rTMS and perceived controllability on pain perception in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age

Exclusion Criteria:

* history of seizures or epilepsy
* family history of seizures
* history of chronic pain conditions
* current depression
* anxiety disorders
* taking any medications shown to lower seizure threshold
* metal implants above the waist
* pregnant
* brain tumors or lesions
* pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Borckardt, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Brain Stimulation Laboratory, Institute of Psychiatry, Charleston, South Carolina, United States

REFERENCES:
- [Result] Borckardt JJ, Reeves ST, Frohman H, Madan A, Jensen MP, Patterson D, Barth K, Smith RA, Gracely R, George MS. Fast left prefrontal rTMS acutely suppresses analgesic effects of perceived controllability on the emotional component of pain experience. Pain. 2011 Jan;152(1):182-187. doi: 10.1016/j.pain.2010.10.018. Epub 2010 Nov 30. PMID 21122992
- See also: Article titled Fast left prefrontal rTMS acutely suppresses analgesic effects of perceived controllability on the emotional component of pain experience — http://www.ncbi.nlm.nih.gov/pubmed/21122992

RESULTS

PARTICIPANT FLOW:
Groups:
- Real TMS: Participants in the real Transcranial Magnetic Stimulation (TMS) group will receive real stimulation across all interventions; the operator role and the receiver role. rTMS will be used to stimulate the left prefrontal cortex using two Neuronetics TMS machines with figure-8, iron core coils at 10Hz and at 110% of resting motor threshold [5 second trains following each trial (25 trials per visit)].
- Sham TMS: Participants in the sham Transcranial Magnetic Stimulation (TMS) group will receive sham stimulation across all interventions; the operator role and the receiver role. Sham Stimulation involves 5 second trains of 10Hz rTMS in pairs alternating between real TMS and eSham TMS (randomly ordered). All sham treatment will be delivered with a specially designed, manufacture-provided sham TMS coil that looks and sounds identical to a real TMS coil but no magnetic current is transferred to the participant.
Period: Overall Study
Arm/Group | Real TMS | Sham TMS
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — failed to experience pain at level 7/10 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real TMS | Sham TMS | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 5 | 6 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Pain Unpleasantness During Perceived Control Condition
Description: The perceived control condtion of the pain task consisted of 30 trials of 1 to 4 seconds of thermal stimulus accompanied by 5 seconds of real or sham TMS). The entire pain task (perceived control condition and no control condition) consisted of 60 trials. Participants in the operator role group rated the unpleasantness of each thermal stimulus on a computerized visual analog scale (VAS). Unpleasantness ratings are on a scale of 0 to 100. 0=not unpleasant. 100=extremely unpleasant. The ratings were averaged over all trials for the perceived control condition for the Real TMS and Sham TMS group. The results below, report the mean unpleasantness rating for both groups during the perceived control condition.
Time Frame: 30 trials of 1 to 4 seconds of thermal stimulus accompanied by 5 seconds of real or sham TMS
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Real TMS | Sham TMS
Number analyzed (Participants) | 12 | 12
units on a scale | 54.5 [48.5 to 59.5] | 60.5 [55.5 to 65.5]

2. Primary Outcome: Pain Intensity During Perceived Control Condition
Description: The perceived control condtion of the pain task consisted of 30 trials of 1 to 4 seconds of thermal stimulus accompanied by 5 seconds of real or sham TMS). The entire pain task (perceived control condition and no control condition) consisted of 60 trials.), participants in the operator role group rated the pain intensity of each thermal stimulus on a computerized visual analog scale (VAS). Pain intensity ratings are on a scale of 0 to 100. 0=not painful. 100=extremely painful. The ratings were averaged over all trials for the perceived control condition for the Real TMS and Sham TMS group. The results below, report the mean pain intensity rating for both groups during the perceived control condition.
Time Frame: 30 trials of 1 to 4 seconds of thermal stimulus accompanied by 5 seconds of real or sham TMS
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Real TMS | Sham TMS
Number analyzed (Participants) | 12 | 12
units on a scale | 51.5 [46 to 56.5] | 57.5 [52.5 to 62.5]

3. Secondary Outcome: Number of Participants That Correctly Guessed Their TMS Condition Assignment
Description: After each participant completed the experiment, they guessed their TMS Condition, whether they received real or sham TMS.
  Results below report the number of participants in each group that guessed their TMS condition correctly.
Time Frame: After Pain Control Paradigm
Measure: Count of Participants; unit: Participants
Arm/Group | Real TMS | Sham TMS
Number analyzed (Participants) | 12 | 12
Participants | 9 | 5
Statistical Analysis 1: Comparison: Real TMS; Test type: Superiority or Other; p = 0.05, Chi-squared; 0.75

4. Secondary Outcome: Confidence Ratings of Guessing TMS Condition Assignment
Description: After participants guessed their TMS condition; whether they received real or sham TMS, They were then asked to rate the confidence in their guess. Ratings were on a scale of 0-10 where 0=complete guess and 10=absolutely sure.
  Results below include the mean confidence ratings of those that guessed the TMS condition correctly and those that guessed incorrectly.
Time Frame: After Pain Control Paradigm
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Correct Guess: 14 of 24 participants guessed the correct TMS condition
- Incorrect Guess: 10/24 participants incorrectly guessed their TMS condition
Arm/Group | Correct Guess | Incorrect Guess
Number analyzed (Participants) | 14 | 10
units on a scale | 5.07 (3.56) | 5.70 (2.83)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Real TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes